CLINICAL TRIAL: NCT05120128
Title: Changes in Inflammatory Biomarkers When Symptomatic Contact Lens Wearers Are Refit in Acuvue Oasys 1-Day Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CR-6433
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: The participant will be masked to the identity of the study lens even though only one arm has been specified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TEST Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers will enter wearing their own lens, then given the TEST Lens for the remainder of the study.
  Interventions: Device: Acuvue® Oasys 1-Day

INTERVENTIONS:
Device: Acuvue® Oasys 1-Day — TEST Lens

SUMMARY:
This is a 5-Visit, single-arm, single-site, subject masked, dispensing trial to evaluate contact lens discomfort and inflammatory biomarker expression.

DETAILED DESCRIPTION:
The study will assess device feasibility for up to 10 habitual wearers of 4 different types of marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 60 (inclusive) years of age at the time of screening.
  4. By self-report, habitually wear one of four soft spherical contact lens types (1-Day Acuvue Moist, Dailies Aqua Comfort Plus, Dailies Total1, Clariti 1 Day) in both eyes in a daily disposable wear modality. Habitual wear is defined as a minimum of 8 hours of wear per day, for a minimum of 4 days per week during the past 4 weeks.
  5. Have a CLDEQ-8 score at pre-screening of 15 or more.
  6. Own a wearable pair of spectacles.
  7. The habitual contact lens sphere correction in each eye must be between -6.00 and -0.50 D or between +0.50 and +4.00 D (inclusive).
  8. The magnitude of the cylinder component of the subject's distance over-refraction must be 1.00 DC or less in each eye.
  9. The subject must have visual acuity of 0.2 high contrast logMAR or better with spherocylinder over-refraction in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or breastfeeding
  2. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See Section 9.1 for additional details regarding excluded systemic medications.
  3. Have had any previous ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, cataract etc.).
  4. Habitually wear multi-focal, toric, or extended wear contact lens correction
  5. Have participated in any contact lens or lens care product clinical trial within 14 days prior to study enrollment
  6. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)
  7. Have a history of amblyopia or strabismus.
  8. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (eg. SynergEyes) within the past 6 months.
  9. Have clinically significant (grade 3 or higher on the Efron grading scale) slit lamp findings (e.g., corneal edema or neovascularization, conjunctival or limbal redness) or any other abnormality which would normally contraindicate contact lens wear
  10. Have any ocular infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
CLDEQ-8 Score follow up 1 | at 1-week follow-up
  Correlation between change in CLDEQ-8 score and change in MMP-9 biomarker expression
CLDEQ-8 Score follow up 2 | at 2-week follow-up
  Correlation between change in CLDEQ-8 score and change in MMP-9 biomarker expression
MMP-9 Expression in Epithelial Cells of Bulbar Conjunctiva | at 1-week follow-up
  Each subject will have EyeprimTM samples collected which involves the 'double impression' technique where samples are collected twice from the same location using a single EyeprimTM membrane. Samples will be collected from the temporal bulbar conjunctiva in both eyes. From these samples, biomarker expression for MMP-9 will be measured. A higher level of MMP-9 expression is associated with a stronger inflammatory response.
MMP-9 Expression in Epithelial Cells of Upper Eyelid Wiper | at 1-week follow-up
  Each subject will have EyeprimTM samples collected which involves the 'double impression' technique where samples are collected twice from the same location using a single EyeprimTM membrane. Samples will be collected from the upper lid margin in both eyes. From these samples, biomarker expression for MMP-9 will be measured. A higher level of MMP-9 expression is associated with a stronger inflammatory response.
MMP-9 Expression in Epithelial Cells of Bulbar Conjunctiva | at 2-week follow-up
  Each subject will have EyeprimTM samples collected which involves the 'double impression' technique where samples are collected twice from the same location using a single EyeprimTM membrane. Samples will be collected from the temporal bulbar conjunctiva in both eyes. From these samples, biomarker expression for MMP-9 will be measured. A higher level of MMP-9 expression is associated with a stronger inflammatory response.
MMP-9 Expression in Epithelial Cells of Upper Eyelid Wiper | at 2-week follow-up
  Each subject will have EyeprimTM samples collected which involves the 'double impression' technique where samples are collected twice from the same location using a single EyeprimTM membrane. Samples will be collected from the upper lid margin in both eyes. From these samples, biomarker expression for MMP-9 will be measured. A higher level of MMP-9 expression is associated with a stronger inflammatory response.

SECONDARY OUTCOMES:
Average difference in CLDEQ-8 scores between Subjects' own lens and AO1D | up to 2-week follow-up
  CLDEQ-8 is a validated outcome measure for soft contact lens wearers. It has been highly correlated with habitual baseline status and change in overall opinion when subjects are refit with contact lenses.10 The sum of the item scores of CLDEQ-8, ranging from 0 to 37, will be used to assess dry eye symptoms, where higher scores indicated more serious symptoms. The score will be calculated for each group (subject's own lens and AO1D) and timepoint (1- and 2-week follow-up). The difference between subjects' own lens and AO1D will be calculated as (AO1D minus subjects' own lens). The average will be reported for each timepoint.
Average Difference in MMP-9 Expression in Epithelial Cells of Bulbar Conjuctiva between Subjects' own lens and AO1D | up to 2 week follow up
  Each subject will have EyeprimTM samples collected which involves the 'double impression' technique where samples are collected twice from the same location using a single EyeprimTM membrane. Samples will be collected from the temporal bulbar conjuctiva in both eyes. From these samples, biomarker expression for MMP-9 will be measured. A higher level of MMP-9 expression is associated with a stronger inflammatory response. The score will be measured for each group (subject's own lens and AO1D) and timepoint (1- and 2-week follow-up). The difference between subjects' own lens and AO1D will be measured as (AO1D minus subjects' own lens). The average difference will be reported for each timepoint.
Average Difference in MMP-9 Expression in Epithelial Cells of Upper Eyelid Wiper between Subjects' own lens and AO1D | up to 2 week follow up
  Each subject will have EyeprimTM samples collected which involves the 'double impression' technique where samples are collected twice from the same location using a single EyeprimTM membrane. Samples will be collected from the upper lid margin in both eyes. From these samples, biomarker expression for MMP-9 will be measured. A higher level of MMP-9 expression is associated with a stronger inflammatory response. The score will be measured for each group (subject's own lens and AO1D) and timepoint (1- and 2-week follow-up). The difference between subjects' own lens and AO1D will be measured as (AO1D minus subjects' own lens). The average difference will be reported for each timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu